CLINICAL TRIAL: NCT02628028
Title: A Randomized, Double-Blind, Placebo-Controlled, 2-Part Phase 2 Study to Evaluate the Safety and Efficacy of LY3337641 in Adult Subjects With Rheumatoid Arthritis: The RAjuvenate Study
Brief Title: A Study of LY3337641 in Rheumatoid Arthritis
Acronym: RAjuvenate
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was terminated after an interim analysis of efficacy and safety data did not warrant continuation of the trial.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16173; I8K-MC-JPDA (Other: Eli Lilly and Company); 2015-003289-97 (EudraCT Number)
Record Dates: First submitted 2015-12-09; First posted 2015-12-11 (Estimated); Results first posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Part A 5 mg LY3337641 (Experimental): Given once a day for 4 weeks.
  Interventions: Drug: LY3337641
- Part A 10 mg LY3337641 (Experimental): Given once a day for 4 weeks.
  Interventions: Drug: LY3337641
- Part A 30 mg LY3337641 (Experimental): Given once a day for 4 weeks.
  Interventions: Drug: LY3337641
- Part A Placebo (Placebo Comparator): Given once a day for 4 weeks.
  Interventions: Drug: Placebo
- Part B 5 mg LY3337641 (Experimental): Given once a day for 12 weeks and an additional 52 weeks for Long-term extension (LTE) period.
  Interventions: Drug: LY3337641
- Part B 10 mg LY3337641 (Experimental): Given once a day for 12 weeks and an additional 52 weeks for Long-term extension (LTE) period.
  Interventions: Drug: LY3337641
- Part B 30 mg LY3337641 (Experimental): Given once a day for 12 weeks and an additional 52 weeks for Long-term extension (LTE) period.
  Interventions: Drug: LY3337641
- Part B Placebo (Placebo Comparator): Given once a day for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3337641 — Administered orally
  Arms: Part A 10 mg LY3337641; Part A 30 mg LY3337641; Part A 5 mg LY3337641; Part B 10 mg LY3337641; Part B 30 mg LY3337641; Part B 5 mg LY3337641
Drug: Placebo — Administered orally
  Arms: Part A Placebo; Part B Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and effectiveness of LY3337641 in adults with rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of childbearing potential test negative for pregnancy at screening and agree not to breastfeed
* Female subjects: agree to use a reliable method of birth control from the start of screening until 28 days after the last dose of study drug or be of nonchildbearing potential
* Male subjects: agree to use a reliable method of birth control from the start of screening until 2 weeks after the last dose of study drug or have undergone vasectomy
* Have a diagnosis of RA based on the 2010 American College of Rheumatology (ACR)/European League against Rheumatism criteria
* Have at least 1 of the following:

  * rheumatoid factor or anti-citrullinated peptide antibodies (ACPA) at screening OR
  * radiographs documenting bony erosions
* Have active RA, defined as:

  * Part A: ≥3 swollen joints (based on 66-joint counts)
  * Part B:
  * ≥6 swollen joints (based on 66-joint counts)
  * ≥6 tender joints (based on 68-joint counts)
  * hsCRP levels greater than the upper limit of normal (ULN) OR positive for ACPA
* Part B only: Have had inadequate response, loss of response, or intolerance to at least 1 synthetic OR biologic disease-modifying antirheumatic drug (DMARD)

Exclusion Criteria:

* Have received any of the following:

  * Part B only: any prior treatment with a product directly targeting Bruton's tyrosine kinase (BTK) (marketed or investigational)
  * belimumab, natalizumab, or vedolizumab within 6 months prior to baseline
  * B-cell-depleting agents (such as rituximab) or other cell-depleting biologics (eg, anti-cluster of differentiation 3 (CD3) antibody) within 12 months prior to screening for Part A or at any time prior to screening for Part B
* Have known hypogammaglobulinemia
* Have hepatitis C virus, hepatitis B virus or human immunodeficiency virus
* Have active tuberculosis (TB)
* Are at high risk of infection or have recent evidence of clinically significant infection
* Have had lymphoma, leukemia, or any malignancy within the previous 5 years except for treated basal cell or squamous epithelial carcinomas of the skin
* Have received a live (attenuated) vaccine within 28 days prior to baseline or plan to receive one during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (60):
- United States (15):
  - Desert Medical Advances, Palm Desert, California
  - Stanford University Hospital, Palo Alto, California
  - Denver Arthritis Center, Denver, Colorado
  - Innovative Research of West Florida, Clearwater, Florida
  - Jeffrey Alper MD Research, Naples, Florida
  - Sun Coast Clinical Research, Inc, New Port Richey, Florida
  - Lovelace Scientific Resources, Venice, Florida
  - Center for Arthritis & Osteoporosis, Elizabethtown, Kentucky
  - Clayton Medical Research, St Louis, Missouri
  - Rowan Regional Medical Center, Salisbury, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Articularis Healthcare d/b/a/ Low Country Rheumatology, PA, North Charleston, South Carolina
  - Accurate Clinical Research, League City, Texas
  - Accurate Clinical Research, Nassau Bay, Texas
  - Rheumatology and Immunotherapy Center, Franklin, Wisconsin
- Argentina (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ciudad Autonoma de Buenos Aire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Fernando
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Miguel de Tucumán
- Australia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maroochydore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Woodville South
- Austria (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Innsbruck
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
- Italy (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torino
- Japan (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Asahikawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kitakyushu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ōmura
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sapporo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sasebo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sendai
- Mexico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Colonia Roma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Distrito Federal
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexicali
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
- Poland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elblag
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nadarzyn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Puerto Rico (3):
  - Office: Perez-De Jesus, Amarilis, Caguas, PR
  - Mindful Medical Research, San Juan, PR
  - Latin Clinical Trial Center, Santurce
- Slovakia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bratislava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zvolen
- South Africa (3):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Pinelands
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stellenbosch
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Umhlanga
- South Korea (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Junggu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alicante
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bilbao
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Seville

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Genovese MC, Spindler A, Sagawa A, Park W, Dudek A, Kivitz A, Chao J, Chan LSM, Witcher J, Barchuk W, Nirula A. Safety and Efficacy of Poseltinib, Bruton's Tyrosine Kinase Inhibitor, in Patients With Rheumatoid Arthritis: A Randomized, Double-blind, Placebo-controlled, 2-part Phase II Study. J Rheumatol. 2021 Jul;48(7):969-976. doi: 10.3899/jrheum.200893. Epub 2020 Dec 15. PMID 33323529
- See also: Click here for more information about this study: A Study of LY3337641 in Participants With Rheumatoid Arthritis (RAjuvenate) — https://lillytrialguide.com/en/studies/rheumatoid-arthritis/JPDA#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consist of 2-parts. Part A included participants with at least mildly active rheumatoid arthritis (RA) and Part B included participants with moderately to severely active RA. Long-term extension (LTE) period allowed eligible participants who completed Part B of study to receive LY3337641 up to an additional 52 weeks.
Groups:
- Part A: Placebo: Participants received oral dose of placebo once daily (QD) for 4 weeks.
- Part A: 5 mg LY3337641: Participants received oral dose of 5 mg LY3337641 QD for 4 weeks.
- Part A: 10 mg LY3337641: Participants received oral dose of 10 mg LY3337641 QD for 4 weeks.
- Part A: 30 mg LY3337641: Participants received oral dose of 30 mg LY3337641 QD for 4 weeks.
- Part B: Placebo: Participants received oral dose of placebo QD for 12 weeks.
- Part B: 5 mg LY3337641: Part B Dosing period: Participants received oral dose of 5 mg LY3337641 tablet QD for 12 weeks.
  Long-term extension (LTE) period: Participants who completed Part B of study received oral dose of 5 mg LY3337641 QD for an additional 52 weeks.
- Part B: 10 mg LY3337641: Participants received oral dose of 10 mg LY3337641 tablet QD for 12 weeks.
  Long-term extension (LTE) period: Participants who completed Part B of study received oral dose of 10 mg LY3337641 QD for an additional 52 weeks.
- Part B: 30 mg LY3337641: Participants received oral dose of 30 mg LY3337641 QD for 12 weeks.
  Long-term extension (LTE) period: Participants who completed Part B of study received oral dose of 30 mg LY3337641 QD for an additional 52 weeks.
Period: Dosing Period
Arm/Group | Part A: Placebo | Part A: 5 mg LY3337641 | Part A: 10 mg LY3337641 | Part A: 30 mg LY3337641 | Part B: Placebo | Part B: 5 mg LY3337641 | Part B: 10 mg LY3337641 | Part B: 30 mg LY3337641
Started | 9 | 9 | 10 | 8 | 62 | 63 | 62 | 63
Received at Least 1dose of Study Drug | 9 | 9 | 10 | 8 | 62 | 63 | 62 | 63
Completed | 9 | 9 | 9 | 8 | 46 | 49 | 46 | 48
Not Completed | 0 | 0 | 1 | 0 | 16 | 14 | 16 | 15
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 2 | 4 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 7 | 6 | 7 | 7
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Site Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 4
Period: Long-term Extension (LTE) Period
Arm/Group | Part A: Placebo | Part A: 5 mg LY3337641 | Part A: 10 mg LY3337641 | Part A: 30 mg LY3337641 | Part B: Placebo | Part B: 5 mg LY3337641 | Part B: 10 mg LY3337641 | Part B: 30 mg LY3337641
Started | 0 (LTE period included participants who completed Part B of the study.) | 0 (LTE period included participants who completed Part B of the study.) | 0 (LTE period included participants who completed Part B of the study.) | 0 (LTE period included participants who completed Part B of the study.) | 0 (Part B LTE was optional;42 participants completed part B placebo period,re-randomized to LTE period.) | 61 (Part B LTE was optional;14 participants completed part B placebo period,re-randomized to LTE period.) | 58 (Part B LTE was optional;14 participants completed part B placebo period,re-randomized to LTE period.) | 61 (Part B LTE was optional;14 participants completed part B placebo period,re-randomized to LTE period.)
Placebo Re-randomized in LTE | 0 | 0 | 0 | 0 | 0 | 14 | 14 | 14
Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 60 | 58 | 61
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 52 | 51 | 51
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 3
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of the study drug.
Groups:
- Part B: 5 mg LY3337641: Participants received oral dose of 5 mg LY3337641 QD for 12 weeks.
- Part B: 10 mg LY3337641: Participants received oral dose of 10 mg LY3337641 QD for 12 weeks.
- Part B: 30 mg LY3337641: Participants received oral dose of 30 mg LY3337641 QD for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo | Part A: 5 mg LY3337641 | Part A: 10 mg LY3337641 | Part A: 30 mg LY3337641 | Part B: Placebo | Part B: 5 mg LY3337641 | Part B: 10 mg LY3337641 | Part B: 30 mg LY3337641 | Total
Number analyzed (Participants) | 9 | 9 | 10 | 8 | 62 | 63 | 62 | 63 | 286
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (11.43) | 54.0 (11.75) | 56.9 (6.44) | 51.9 (5.72) | 50.5 (8.75) | 50.1 (9.20) | 51.7 (9.36) | 51.9 (8.91) | 51.5 (9.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 9 | 5 | 54 | 53 | 56 | 53 | 246
  Male | 1 | 1 | 1 | 3 | 8 | 10 | 6 | 10 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 3 | 2 | 34 | 26 | 23 | 21 | 116
  Not Hispanic or Latino | 5 | 6 | 7 | 6 | 24 | 29 | 26 | 23 | 126
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 4 | 8 | 13 | 19 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 6
  Asian | 0 | 0 | 0 | 0 | 7 | 14 | 9 | 10 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 1 | 1 | 2 | 2 | 2 | 10
  White | 6 | 7 | 9 | 7 | 53 | 46 | 50 | 51 | 229
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 0 | 0 | 0 | 0 | 4 | 2 | 3 | 5 | 14
  Argentina | 0 | 0 | 0 | 0 | 15 | 13 | 15 | 14 | 57
  United States | 6 | 6 | 6 | 7 | 12 | 13 | 15 | 6 | 71
  Japan | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 7 | 25
  Spain | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 6 | 13
  South Korea | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 3 | 8
  Austria | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Poland | 0 | 0 | 2 | 1 | 9 | 9 | 4 | 7 | 32
  Italy | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 5 | 10
  Mexico | 3 | 3 | 2 | 0 | 10 | 6 | 7 | 4 | 35
  South Africa | 0 | 0 | 0 | 0 | 2 | 3 | 5 | 3 | 13
  Slovakia | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4
  Australia | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Treatment-Emergent Adverse Events (TEAEs) or Adverse Events of Special Interest (AESIs) or Any Serious AEs (SAEs) in Part A
Description: TEAEs are any untoward medical occurrence that either occurs or worsens at any time after treatment baseline, and in the opinion of the investigators is possibly related to study drug. Skin Rash was the only event that was considered an AESI. A serious AE is defined as an event that results in death, initial or prolonged hospitalization, is life-threatening, leads to persistent or significant disability/incapacity, is associated with congenital anomaly/birth defect, or is considered significant by the investigator for any other reason. A summary of SAEs and other non-serious AEs, regardless of whether or not they were possibly related to study drug, is located in the Reported Adverse Event section.
Time Frame: Up to 6 Weeks
Population: All randomized participants who received at least 1 dose of the study drug in Part A.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: 5 mg LY3337641 | Part A: 10 mg LY3337641 | Part A: 30 mg LY3337641
Number analyzed (Participants) | 9 | 9 | 10 | 8
Participants
  TEAEs | 3 | 1 | 6 | 2
  AESIs | 0 | 0 | 0 | 0
  SAEs | 0 | 0 | 0 | 0

2. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response in Part B
Description: ACR20 Responder Index is a composite of clinical, laboratory, and functional measures in rheumatoid arthritis (RA). "ACR20 Responder" is a participant who has at least 20% improvement in both tender and swollen joint counts and in at least 3 of the following 5 criteria: Physician's Global Assessment of Disease Activity, Patient's Global Assessment of Disease Activity, Patient's Global Assessment of Arthritis Pain using visual analog scale (VAS), Health Assessment Questionnaire - Disability Index (HAQ-DI) and high-sensitivity C-reactive protein (hsCRP). Participants with missing responses and /or participants who discontinue study or drug before analysis timepoint are deemed non-responders.
Time Frame: Week 12
Population: All randomized participants who received at least 1 dose of the study drug, for participants who completed or early discontinued dosing treatment period before the study was terminated in Part B. Missing values due to discontinuation of study or drug, or missing data were imputed using non-responder imputation (NRI).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part B: Placebo | Part B: 5 mg LY3337641 | Part B: 10 mg LY3337641 | Part B: 30 mg LY3337641
Number analyzed (Participants) | 54 | 56 | 52 | 55
Percentage of Participants | 48.1 [34.8 to 61.5] | 55.4 [42.3 to 68.4] | 44.2 [30.7 to 57.7] | 50.9 [37.7 to 64.1]
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: 5 mg LY3337641; Test type: Superiority; p = 0.473, Regression, Logistic
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: 10 mg LY3337641; Test type: Superiority; p = 0.670, Regression, Logistic
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: 30 mg LY3337641; Test type: Superiority; p = 0.823, Regression, Logistic

3. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response in Part B
Description: ACR50 Responder Index is composite of clinical, laboratory, and functional measures in RA. "ACR50 Responder" is a participant who has at least 50% improvement in both tender and swollen joint counts and in at least 3 of the following 5 criteria:
  Physician's Global Assessment of Disease Activity, Patient's Global Assessment of Disease Activity, Patient's Global Assessment of Arthritis Pain using VAS, HAQ-DI and hsCRP. Participants with missing responses and/or participants who discontinue study or drug before analysis timepoint are deemed non-responders.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part B: Placebo | Part B: 5 mg LY3337641 | Part B: 10 mg LY3337641 | Part B: 30 mg LY3337641
Number analyzed (Participants) | 54 | 56 | 52 | 55
Percentage of Participants | 27.8 [15.8 to 39.7] | 25.0 [13.7 to 36.3] | 15.4 [5.6 to 25.2] | 29.1 [17.1 to 41.1]
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: 5 mg LY3337641; Test type: Superiority; p = 0.743, Regression, Logistic
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: 10 mg LY3337641; Test type: Superiority; p = 0.124, Regression, Logistic
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: 30 mg LY3337641; Test type: Superiority; p = 0.858, Regression, Logistic

4. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response in Part B
Description: ACR70 Responder Index is composite of clinical, laboratory, and functional measures in RA. "ACR70 Responder" is a participant who has at least 70% improvement in both tender and swollen joint counts and in at least 3 of the following 5 criteria:
  Physician's Global Assessment of Disease Activity, Patient's Global Assessment of Disease Activity, Patient's Global Assessment of Arthritis Pain using VAS, HAQ-DI and hsCRP. Participants with missing responses and/or participants who discontinue study or drug before analysis timepoint are deemed non-responders.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part B: Placebo | Part B: 5 mg LY3337641 | Part B: 10 mg LY3337641 | Part B: 30 mg LY3337641
Number analyzed (Participants) | 54 | 56 | 52 | 55
Percentage of Participants | 16.7 [6.7 to 26.6] | 8.9 [1.5 to 16.4] | 1.9 [0.0 to 5.7] | 16.4 [6.6 to 26.1]
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: 5 mg LY3337641; Test type: Superiority; p = 0.199, Regression, Logistic
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: 10 mg LY3337641; Test type: Superiority; p = 0.028, Regression, Logistic
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: 30 mg LY3337641; Test type: Superiority; p = 0.863, Regression, Logistic

5. Secondary Outcome: Change From Baseline in the Disease Activity Score (DAS) 28-high-sensitivity C-reactive Protein (hsCRP) in Part B
Description: Disease Activity Score (DAS) modified to include 28 joint count (DAS28) consisted of composite score of following variables: tender joint count (TJC28), swollen joint count (SJC28), C-reactive protein (CRP) (milligrams per liter), and Patient's Global Assessment of Disease Activity using VAS. DAS28 was calculated using following formula: DAS28-CRP=0.56*square root (sqrt)(TJC28)+0.28*sqrt(SJC28)+0.36*natural log(CRP+1)+0.014*Patient's Global VAS+0.96. Scores ranged 1.0-9.4, where lower scores indicated less disease activity.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part B: Placebo | Part B: 5 mg LY3337641 | Part B: 10 mg LY3337641 | Part B: 30 mg LY3337641
Number analyzed (Participants) | 62 | 63 | 62 | 63
units on a scale | -1.62 (1.447) | -1.55 (1.182) | -1.24 (1.146) | -1.80 (1.453)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: 5 mg LY3337641; Test type: Superiority; p = 0.863, Mixed-effects Model for Repeated Measure; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.53 to 0.44], Standard Error of Mean 0.25
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: 10 mg LY3337641; Test type: Superiority; p = 0.503, Mixed-effects Model for Repeated Measure; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.32 to 0.65], Standard Error of Mean 0.25
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: 30 mg LY3337641; Test type: Superiority; p = 0.289, Mixed-effects Model for Repeated Measure; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.77 to 0.23], Standard Error of Mean 0.25

6. Secondary Outcome: Percentage of Participants Who Achieve Low Disease Activity Using DAS28-hsCRP in Part B
Description: as for outcome 5
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part B: Placebo | Part B: 5 mg LY3337641 | Part B: 10 mg LY3337641 | Part B: 30 mg LY3337641
Number analyzed (Participants) | 54 | 56 | 52 | 55
Percentage of Participants | 27.8 [15.8 to 39.7] | 32.1 [19.9 to 44.4] | 21.2 [10.1 to 32.3] | 29.1 [17.1 to 41.1]
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: 5 mg LY3337641; Test type: Superiority; p = 0.626, Regression, Logistic
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: 10 mg LY3337641; Test type: Superiority; p = 0.418, Regression, Logistic
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: 30 mg LY3337641; Test type: Superiority; p = 0.951, Regression, Logistic

7. Secondary Outcome: Percentage of Participants Who Achieve Clinical Remission Using DAS28-hsCRP in Part B
Description: Disease Activity Score (DAS) modified to include 28 joint count (DAS28) consisted of composite score of following variables: tender joint count (TJC28), swollen joint count (SJC28), C-reactive protein (CRP) (milligrams per liter), and Patient's Global Assessment of Disease Activity using visual analog scale (VAS) (participant global VAS). DAS28 was calculated using following formula: DAS28-CRP=0.56*square root (sqrt)(TJC28)+0.28*sqrt(SJC28)+0.36*natural log(CRP+1)+0.014*Patient's Global VAS+0.96. Clinical remission is defined as DAS28-hsCRP <2.6.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part B: Placebo | Part B: 5 mg LY3337641 | Part B: 10 mg LY3337641 | Part B: 30 mg LY3337641
Number analyzed (Participants) | 54 | 56 | 52 | 55
Percentage of Participants | 20.4 [9.6 to 31.1] | 19.6 [9.2 to 30.0] | 7.7 [0.4 to 14.9] | 25.5 [13.9 to 37.0]
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: 5 mg LY3337641; Test type: Superiority; p = 0.905, Regression, Logistic
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: 10 mg LY3337641; Test type: Superiority; p = 0.069, Regression, Logistic
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: 30 mg LY3337641; Test type: Superiority; p = 0.547, Regression, Logistic

8. Secondary Outcome: Pharmacokinetics (PK): Clearance Parameter of LY3337641
Description: Apparent total body clearance of drug after oral administration based on population PK analysis was evaluated. As prespecified per protocol, an overall population estimate of clearance is generated and data from Part A and B were combined for the analysis. The sparse data was then analyzed using population PK methods in Non linear Mixed Effects Model (NONMEM) to generate an overall population estimate of clearance.
Time Frame: Part A: Weeks 1, 2, and 4, Day 1 (0.5 to 2 hours postdose); Part B: Weeks 2, 4, 8, and 12, Day 1 (0.5 to 2 hours postdose)
Population: All randomized participants who received at least 1 dose of the study drug and have evaluable PK data in in Part A and Part B.
Measure: Mean (Standard Error); unit: Liter per hour (L/hr)
Groups:
- LY3337641: Participants received oral doses of 5 mg, 10 mg and 30 mg LY3337641 QD for 4 weeks in Part A and 12 weeks in Part B.
Arm/Group | LY3337641
Number analyzed (Participants) | 209
Liter per hour (L/hr) | 29.1 (5.9)

ADVERSE EVENTS:
Time Frame: Up to 88 Weeks
Description: All randomized participants who received at least 1 dose of the study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Long-Term Extension: 5 mg LY3337641: Participants who completed Part B of study received oral dose of 5 mg LY3337641 QD for an additional 52 weeks.
- Long-Term Extension: 10 mg LY3337641: Participants who completed Part B of study received oral dose of 10 mg LY3337641 QD for an additional 52 weeks.
- Long-Term Extension: 30 mg LY3337641: Participants who completed Part B of study received oral dose of 30 mg LY3337641 QD for an additional 52 weeks.
Arm/Group | Part A: Placebo | Part A: 5 mg LY3337641 | Part A: 10 mg LY3337641 | Part A: 30 mg LY3337641 | Part B: Placebo | Part B: 5 mg LY3337641 | Part B: 10 mg LY3337641 | Part B: 30 mg LY3337641 | Long-Term Extension: 5 mg LY3337641 | Long-Term Extension: 10 mg LY3337641 | Long-Term Extension: 30 mg LY3337641
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/10 | 0/8 | 0/62 | 0/63 | 0/62 | 1/63 | 0/61 | 0/58 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/10 | 0/8 | 2/62 | 0/63 | 0/62 | 3/63 | 1/61 | 3/58 | 1/61
Other Adverse Events (participants affected / at risk) | 3/9 | 1/9 | 6/10 | 2/8 | 7/62 | 10/63 | 12/62 | 19/63 | 11/61 | 12/58 | 10/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo (N=9) | Part A: 5 mg LY3337641 (N=9) | Part A: 10 mg LY3337641 (N=10) | Part A: 30 mg LY3337641 (N=8) | Part B: Placebo (N=62) | Part B: 5 mg LY3337641 (N=63) | Part B: 10 mg LY3337641 (N=62) | Part B: 30 mg LY3337641 (N=63) | Long-Term Extension: 5 mg LY3337641 (N=61) | Long-Term Extension: 10 mg LY3337641 (N=58) | Long-Term Extension: 30 mg LY3337641 (N=61)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part A: Placebo (N=9) | Part A: 5 mg LY3337641 (N=9) | Part A: 10 mg LY3337641 (N=10) | Part A: 30 mg LY3337641 (N=8) | Part B: Placebo (N=62) | Part B: 5 mg LY3337641 (N=63) | Part B: 10 mg LY3337641 (N=62) | Part B: 30 mg LY3337641 (N=63) | Long-Term Extension: 5 mg LY3337641 (N=61) | Long-Term Extension: 10 mg LY3337641 (N=58) | Long-Term Extension: 30 mg LY3337641 (N=61)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (4) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (2) | 5 (5) | 1 (1) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (4) | 4 (4)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 4 (4) | 2 (2) | 1 (1) | 1 (2) | 2 (2)
Carotid artery aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/1 (0) | 0/1 (0) | 0/1 (0) | 0/3 (0) | 1/8 (1) | 0/10 (0) | 0/6 (0) | 0/10 (0) | 0/9 (0) | 0/4 (0) | 0/10 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0/1 (0) | 0/1 (0) | 0/1 (0) | 0/3 (0) | 0/8 (0) | 0/10 (0) | 0/6 (0) | 1/10 (1) | 0/9 (0) | 0/4 (0) | 0/10 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
The trial was terminated after an interim analysis of efficacy and safety data did not warrant continuation of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/28/NCT02628028/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT02628028/SAP_001.pdf